CLINICAL TRIAL: NCT00760903
Title: Magnetic Resonance (MR) Spectroscopy and Diffusion Tensor Imaging in Determining Brain Injury and Subsequent Clinical Outcome in Patients of Moderate Brain Trauma
Status: Withdrawn | Type: Observational
Why Stopped: Study was not started due to PI concentrating on other studies
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Pia C Maly Sundgren, MD, PhD, Principal Investigator, University of Michigan
Other Study IDs: 2003-0053
Record Dates: First submitted 2008-09-24; First posted 2008-09-26 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Brain Trauma
Keywords: Moderate brain trauma
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- > 18 years moderate head trauma: Group I: (Pilot group): 5-10 patients > 18 years old, gender and race indifferent with moderate head trauma.
  Interventions: Other: Conventional MRI of the brain; Other: MR spectroscopy (MRS); Other: MR Diffusion Tensor Imaging (DTI)
- > 18, gender and race indifferent: Group II: 30 patients > 18 years old, gender, and race indifferent with moderate head trauma
  Interventions: Other: Conventional MRI of the brain; Other: MR spectroscopy (MRS); Other: MR Diffusion Tensor Imaging (DTI)
- Pediatric: Group III: 30 patients < 18 years old, gender and race indifferent with moderate head trauma (pediatric patient group)
  Interventions: Other: Conventional MRI of the brain; Other: MR spectroscopy (MRS); Other: MR Diffusion Tensor Imaging (DTI)
- Pre-evaluated: Group IV: 10-20 patients age, gender and race indifferent with moderate head trauma that have been examined with conventional MRI of the brain, MRS and DTI as clinically requested. The images of these patients will be evaluated retrospectively for data- point collection.
  Interventions: Other: Conventional MRI of the brain; Other: MR spectroscopy (MRS); Other: MR Diffusion Tensor Imaging (DTI)
- Control Group: Group V (control group): 20 volunteers without prior history of traumatic brain injury or neurological problems.
  Interventions: Other: Conventional MRI of the brain; Other: MR spectroscopy (MRS); Other: MR Diffusion Tensor Imaging (DTI)

INTERVENTIONS:
Other: Conventional MRI of the brain
Other: MR spectroscopy (MRS)
Other: MR Diffusion Tensor Imaging (DTI)

SUMMARY:
The purpose of this study is to use magnetic resonance spectroscopy (MRS) and diffusion tensor imaging (DTI) to assess for traumatic brain injury and determine if there is any correlation of these findings to clinical outcome. MR spectroscopy using 2D-CSI (a multi voxel technique) of the corpus callosum, basal ganglia, lobar white matter and brainstem may reveal areas of injury and quantification of the metabolites from these areas may be used to correlate with imaging findings and clinical evaluation. White matter disruption in these areas is commonly seen after TBI, caused by diffuse axonal injury. It has been implicated in the long term outcomes in these patients, but has been difficult to assess by standard radiologic studies.

By the use of DTI it may be possible to demonstrate damaged white matter tracts which could be helpful in the evaluation of traumatic brain injury. Most TBI subjects have injuries that involved torque to the brain. This results in a shearing injury to the long white matter tracts, which has been hypothesized to be related to cognitive outcome.

Also, to demonstrate that MRS and DTI prove valuable in predicting outcome in patients of moderate brain trauma by conducting progressive studies acutely (within 24 hours) and long term (4-6 weeks). Most patients will most likely be followed clinically for over a year, and, if clinical indicated, farther scanning can be done at a later date.

By comparing fraction anisotropy, ADC values, and metabolic ratios by the use of DTI and MRS in the adult and pediatric populations, may help to assess differences in recovery.

Lastly, a comparison between the two groups in changes in brain metabolism and/or white matter tract disruption/re-connection after TBI with and/or without links to outcome can be done.

DETAILED DESCRIPTION:
The purpose of this study is to determine if MRI imaging can accurately detect the clinical outcome (extent of recovery) of patients who have moderate to severe brain injury. This study may show that MRI can provide a clearer picture on the extent of the brain injury and help medical physicians decide how to best treat these patients with a more accurate idea of the brain function of the recovering patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients of acute moderate brain trauma

Exclusion Criteria:

* Patients who are medically unstable or have CT findings that may interfere with the study such as:

  * a large hemorrhage or edema
  * encephalomalacia
  * prior neurosurgeries
  * hardware placed in the head or neck
  * prior head trauma
  * history of neurological conditions

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Have had a clinically ordered CT exam performed within 24 hours of admission to the hospital. We will be enrolling 5 different groups of subjects into this study. These groups include patients18 years of age or older with moderate to severe head trauma. Children under 18 years of age with moderate to severe head trauma. A group of patients of any age who have already undergone conventional MRI of the brain and a group of volunteers who are part of another research study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2003-06; Primary Completion 2008-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To determine if MRI imaging can accurately detect the clinical outcome (extent of recovery) of patients who have moderate to severe brain injury. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No